CLINICAL TRIAL: NCT02684279
Title: An Open-label, Flexibly-dosed, Multicenter, Extension Study of Dasotraline to Evaluate Long-term Safety and Tolerability in Adults With Binge-eating Disorder
Brief Title: Dasotraline Binge Eating Disorder Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEP360-322
Record Dates: First submitted 2016-01-28; First posted 2016-02-17 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Binge Eating Disorder
MeSH Terms: conditions — Binge-Eating Disorder | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine

STUDY DESIGN:
Masking Description: open-label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dasotraline (Experimental): 4, 6, 8 mg flexibly dosed
  Interventions: Drug: Dasotraline

INTERVENTIONS:
Drug: Dasotraline — Dasotraline 4, 6, 8 mg flexibly dosed once daily

SUMMARY:
Binge Eating Disorder Extension Study.

DETAILED DESCRIPTION:
This is a Phase 3, 12 month, multicenter, open-label, flexibly-dosed, safety study in adults with Binge Eating Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the treatment period of a dasotraline core study (ie, SEP360 221 or SEP360-321) for the treatment of BED.
* Subject has agreed to participate by providing written informed consent and is willing and able to comply with the protocol, in the opinion of the investigator.
* Subject has not taken any medication other than the study drug for the purpose of controlling BED symptoms during the core study.
* Female subject must have a negative urine pregnancy test at open label (OL) Baseline; females who are post-menopausal (defined as at least 12 months of spontaneous amenorrhea) and those who have undergone hysterectomy or bilateral oophorectomy will be exempted from the pregnancy test.
* Female subject of childbearing potential and male subject with female partner of childbearing potential must agree to use an effective and medically acceptable form of birth control (see Section 22, Appendix III) throughout the study period. Note: Continued use of an effective and medically acceptable form of birth control is recommended for 30 days after study completion.
* Subject is judged by the investigator to be suitable for participation in a 12 month clinical trial involving open-label dasotraline treatment.
* Subject can read well enough to understand the informed consent form and other subject materials.

Exclusion Criteria:

* Subject is considered by the investigator to be at imminent risk of suicide, injury to self or to others, or damage to property.
* Subject is considered a suicide risk in the investigator's opinion or has any previous history of suicide attempt within the past 12 months.
* Subject answers "yes" to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C SSRS assessment at OL Baseline. Subjects who answer "yes" to this question must be referred to the Investigator for follow up evaluation.
* Subject has a clinically significant abnormality including physical examination, vital signs, ECG, or laboratory tests that the investigator in consultation with the medical monitor considers to be inappropriate to allow participation in the study.
* Subject has a positive urine drug screen (UDS) or breath alcohol test at OL Baseline.
* Subject is breastfeeding.
* Subject is at high risk of non-compliance in the investigator's opinion.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 533 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dasotraline Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (57):
- United States (57):
  - Noesis Parma, Phoenix, Arizona
  - Southern California Research, Beverly Hills, California
  - Pharmacology Research Institute, Encino, California
  - Collaborative NeuroScience Network Inc., Garden Grove, California
  - Pharmacology Research Institute, Newport Beach, California
  - Artemis Institute for Clinical Research, San Marcos, California
  - Syrentis Clinical Research, Santa Ana, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Weiss and Lytle, PLLC, Denver, Colorado
  - CT Clinical Research, Cromwell, Connecticut
  - Gulfcoast Clinical Research Center, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Miami Research Associates, South Miami, Florida
  - Institute of Advanced Medical Research, Alpharetta, Georgia
  - Neuotrials Research, Inc., Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Capstone Clinical Research, Libertyville, Illinois
  - Goldpoint Clinical Research, Inc., Indianapolis, Indiana
  - Phoenix Medical Research, Inc. Suite 135, Prairie Village, Kansas
  - Cyress Medical Research Center, LLC, Wichita, Kansas
  - McLean Hospital, Belmont, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - ActivMed Practices & Research, Inc., Methuen, Massachusetts
  - Adams Clinical Trials, LLC, Watertown, Massachusetts
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - ActivMed Practices and Research, Inc., Portsmouth, New Hampshire
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Princeton Medical Institute, LCC, Princeton, New Jersey
  - Bioscience Research, LLC, Mount Kisco, New York
  - Manhattan Behavioral Medicine, PLLC, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Wake Research Associates, Raleigh, North Carolina
  - Radiant Research, Inc., Akron, Ohio
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Lindner Center Of Hope, Mason, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Oregon Center for Clinical Investigatons, INC., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Lehigh Center For Clinical Research, Allentown, Pennsylvania
  - Radiant Research, Inc., Anderson, South Carolina
  - Radient Research, Inc., Greer, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - Clinical Neuroscience Solutons, Inc., Memphis, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Donald J. Garcia Jr., MD, Austin, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Psychiatric Medical Associates, Plano, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radient Research, Inc., San Antonio, Texas
  - Radiant Research, Inc., Murray, Utah
  - Neuropsychiatric Associates, Woodstock, Vermont
  - NeuroScience, Inc., Herndon, Virginia
  - Summitt Research Network(Seattle) LLC, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 533 subjects were enrolled in this study. Five subjects did not receive any dose of study medication.
Period: Overall Study
Arm/Group | Dasotraline
Started | 528
Completed | 249
Not Completed | 279
Not completed — Adverse Event | 87
Not completed — Lack of Efficacy | 4
Not completed — Lost to Follow-up | 61
Not completed — Protocol Violation | 6
Not completed — Pregnancy | 8
Not completed — Withdrawal by Subject | 92
Not completed — non-compliance with study drug | 9
Not completed — non compliance with study visits | 2
Not completed — subject to have surgery | 1
Not completed — family emergency | 1
Not completed — Site closures | 7
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: safety
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 526
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.8 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 440
  Male | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 85
  Not Hispanic or Latino | 443
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 82
  White | 420
  More than one race | 11
  Unknown or Not Reported | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 167.4 (8.77)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 95.1 (21.52)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 33.8 (6.348)
Binge-eating Clinical Global Impression-Severity (BE-CGI-S) Score at Double-Blind (DB) Baseline [Mean (Standard Deviation); unit: Score] — DB Baseline (ie, Baseline assessment of the double-blind core studies [SEP 360-221, or SEP360-321]) is defined as the last assessment made on or before the 1st dose of double-blind study medication as described in the SAPs of the core studies.
  Score | 4.5 (0.54)
Binge-eating Clinical Global Impression-Severity (BE-CGI-S) Score at Open Label (OL) Baseline [Mean (Standard Deviation); unit: Score] — The OL Baseline is defined as the last assessment made on or before Day 1 of the extension study (ie, Baseline assessment in the open-label study [SEP 360-322] for demographic and EDE-Q modified, and height at the screening and the Endpoint assessment of the double-blind studies [SEP 360-221, or SEP 360-321], otherwise).
  Score | 2.4 (1.38)
Eating Disorder Examination Question(EDE-QM) Modified Score at DB Baseline - Global Score [Mean (Standard Deviation); unit: Score] — DB Baseline (ie, Baseline assessment of the double-blind core studies [SEP 360-221, or SEP360-321]) is defined as the last assessment made on or before the 1st dose of double-blind study medication as described in the SAPs of the core studies.
  Score | 3.7 (1.522)
Eating Disorder Examination Question(EDE-QM) Modified Score at DB Baseline - Restraint [Mean (Standard Deviation); unit: Score] — DB Baseline (ie, Baseline assessment of the double-blind core studies [SEP 360-221, or SEP360-321]) is defined as the last assessment made on or before the 1st dose of double-blind study medication as described in the SAPs of the core studies.
  Score | 2.21 (2.007)
Eating Disorder Examination Question(EDE-QM) Modified Score at DB Baseline - Shape Concern [Mean (Standard Deviation); unit: Score] — DB Baseline (ie, Baseline assessment of the double-blind core studies [SEP 360-221, or SEP360-321]) is defined as the last assessment made on or before the 1st dose of double-blind study medication as described in the SAPs of the core studies.
  Score | 4.38 (1.721)
EDE-QM Modified Score at DB Baseline - Weight Concern [Mean (Standard Deviation); unit: Score] — DB Baseline (ie, Baseline assessment of the double-blind core studies [SEP 360-221, or SEP360-321]) is defined as the last assessment made on or before the 1st dose of double-blind study medication as described in the SAPs of the core studies.
  Score | 4.5 (1.655)
EDE-QM Modified Score at OL Baseline - Global Score [Mean (Standard Deviation); unit: Score] — The OL Baseline is defined as the last assessment made on or before Day 1 of the extension study (ie, Baseline assessment in the open-label study [SEP 360-322] for demographic and EDE-Q modified, and height at the screening and the Endpoint assessment of the double-blind studies [SEP 360-221, or SEP 360-321], otherwise).
  Score | 2.9 (1.687)
EDE-QM Modified Score at OL Baseline - Restraint [Mean (Standard Deviation); unit: Score] — The OL Baseline is defined as the last assessment made on or before Day 1 of the extension study (ie, Baseline assessment in the open-label study [SEP 360-322] for demographic and EDE-Q modified, and height at the screening and the Endpoint assessment of the double-blind studies [SEP 360-221, or SEP 360-321], otherwise).
  Score | 1.71 (1.961)
EDE-QM Modified Score at OL Baseline - Shape Concern [Mean (Standard Deviation); unit: Score] — The OL Baseline is defined as the last assessment made on or before Day 1 of the extension study (ie, Baseline assessment in the open-label study [SEP 360-322] for demographic and EDE-Q modified, and height at the screening and the Endpoint assessment of the double-blind studies [SEP 360-221, or SEP 360-321], otherwise).
  Score | 3.44 (1.944)
Eating Disorder Examination Question(EDE-QM) Modified Score at OL Baseline - Weight Concern [Mean (Standard Deviation); unit: Score] — The OL Baseline is defined as the last assessment made on or before Day 1 of the extension study (ie, Baseline assessment in the open-label study [SEP 360-322] for demographic and EDE-Q modified, and height at the screening and the Endpoint assessment of the double-blind studies [SEP 360-221, or SEP 360-321], otherwise).
  Score | 3.55 (1.912)
summary for Body Mass Index (BMI) category at open label baseline [Count of Participants; unit: Participants] — The OL Baseline is defined as the last assessment made on or before Day 1 of the extension study (ie, Baseline assessment in the open-label study [SEP 360-322] for demographic and EDE-Q modified, and height at the screening and the Endpoint assessment of the double-blind studies [SEP 360-221, or SEP 360-321], otherwise).
  Participants
    Underweight/Normal (<25) | 53
    Overweight (25 to <30) | 104
    Obesity Class I (30 to <35) | 134
    Obesity Class II (35 to <40) | 136
    Obesity Class III (>=40) | 101

OUTCOME MEASURES:

1. Primary Outcome: Frequency and Severity of Suicidal Ideation Using the Columbia-suicide Severity Rating Scale (C-SSRS)
Description: Columbia-suicide severity rating scale (C-SSRS) Severity of suicidal ideation is rated on a 6-point scale from 0='No ideation present' to 5='Active ideation with plan and intent'. A score of 4 or 5 on this scale indicates serious suicidal ideation. Suicidal behavior is collected as presence/absence of actual attempts, non-suicidal self-injurious behavior, interrupted attempts, aborted attempts, preparatory acts or behavior, and any suicidal behavior
Time Frame: Baseline to Week 52
Population: Safety- please note:
  one subject had no value for Suicidal Ideation or Suicidal Behavior
Measure: Count of Participants; unit: Participants
Arm/Group | Dasotraline
Number analyzed (Participants) | 527
Participants
  0: No suicidal ideation | 515
  1: Wish to be dead | 7
  2: Non-specific active suicidal thoughts | 3
  3: ideation with any methods , no intent to act | 1
  4: ideation with some intent to act, no plan | 0
  5: Active ideation with specific plan and intent | 1

2. Primary Outcome: Frequency and Severity of Suicidal Behavior Using the C-SSRS
Description: as for outcome 1
Time Frame: Baseline to Week 52
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Dasotraline
Number analyzed (Participants) | 527
Participants
  Preparatory acts or behavior | 1
  Aborted attempt | 0
  Interrupted attempt | 0
  Actual attempt | 1
  Completed suicide | 0

3. Secondary Outcome: Change in Body Weight
Description: Change in body weight
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
kg
  Change from DB Baseline Week 52 Endpoint | -4.65 [-5.36 to -3.93]
  Change from OL Baseline Week 52 Endpoint | -2.13 [-2.77 to -1.49]

4. Secondary Outcome: Percent Change in Body Weight (kg)
Description: Percent change in body weight (kg)
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
percent change
  % Change from DB Baseline Week 52 Endpoint | -4.65 [-5.35 to -3.95]
  % Change from OL Baseline Week 52 Endpoint | -2.07 [-2.71 to -1.43]

5. Secondary Outcome: Change in Body Mass Index
Description: Change in Body Mass Index
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
kg/m^2
  Change from DB Baseline Week 52 Endpoint | -1.64 [-1.89 to -1.39]
  Change from OL Baseline Week 52 Endpoint | -0.75 [-0.97 to -0.53]

6. Secondary Outcome: Percent Change in Body Mass Index (kg/m^2)
Description: Percent change in Body Mass Index (kg/m^2)
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
percent change
  % Change from DB Baseline Week 52 Endpoint | -4.65 [-5.35 to -3.95]
  % Change from OL Baseline Week 52 Endpoint | -2.07 [-2.71 to -1.43]

7. Secondary Outcome: Change in Fasting Lipid Panel, Triglyceride's
Description: Change in fasting lipid panel, Triglyceride's
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
mg/dL
  Change from DB Baseline Week 52 Endpoint | -11.9 [-17.5 to -6.3]
  Change from OL Baseline Week 52 Endpoint | -5.3 [-10.4 to -0.3]

8. Secondary Outcome: Change in Fasting Lipid Panel , Total Cholesterol
Description: Change in fasting lipid panel , total cholesterol
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
mg/dL
  Change from DB Baseline Week 52 Endpoint | -7.0 [-9.3 to -4.8]
  Change from OL Baseline Week 52 Endpoint | -3.5 [-5.6 to -1.4]

9. Secondary Outcome: Change in Fasting Lipid Panel , High-density Lipoprotein [HDL] Cholesterol,
Description: Change in fasting lipid panel, high-density lipoprotein [HDL] cholesterol,
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
mg/dL
  Change from DB Baseline Week 52 Endpoint | -1.1 [-2.0 to -0.2]
  Change from OL Baseline Week 52 Endpoint | 1.1 [0.2 to 1.9]

10. Secondary Outcome: Change in Fasting Lipid Panel, Low-density Lipoprotein [LDL] Cholesterol)
Description: Change in fasting lipid panel, low-density lipoprotein [LDL] cholesterol)
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
mg/dL
  Change from DB Baseline Week 52 Endpoint | -3.6 [-5.5 to -1.6]
  Change from OL Baseline Week 52 Endpoint | -3.4 [-5.2 to -1.5]

11. Secondary Outcome: Change in Hemoglobin A1c Levels
Description: Change in hemoglobin A1c levels
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
Percent change
  Change from DB Baseline Week 52 Endpoint | 0.00 [-0.02 to 0.02]
  Change from OL Baseline Week 52 Endpoint | 0.00 [-0.02 to 0.02]

12. Secondary Outcome: Change in Fasting Glucose Levels
Description: Change in fasting glucose levels
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
mg/dL
  Change from DB Baseline Week 52 Endpoint | 2.2 [0.9 to 3.5]
  Change from OL Baseline Week 52 Endpoint | 1.7 [0.3 to 3.1]

13. Secondary Outcome: Change in Eating Disorder Examination Questionnaire (EDE Q) Modified Global Score and Subscale Scores (Restraint, Shape, Concern, Weight Concern), and Items 4-6 Scores
Description: Eating Disorder Examination Questionnaire (EDE-Q) Modified global and subscale scores 4 subscale scores (Restraint, Eating Concern, Shape Concern, and Weight Concern) range from 0- 6, where 0 represents absence of the feature and 6 represents an extreme degree. An EDE-Q global score is calculated as average of 4 EDE-Q subscale scores.
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
units on a scale
  Global Score Change from DB Baseline Endpoint | -1.16 [-1.30 to -1.02]
  Global Score Change from OL Baseline Endpoint | -0.37 [-0.48 to -0.26]
  Restraint Change from DB Baseline Endpoint | -0.63 [-0.81 to -0.45]
  Restraint Change from OL Baseline Endpoint | -0.13 [-0.27 to 0.01]
  Shape Concern Change from DB Baseline Endpoint | -1.38 [-1.54 to -1.22]
  Shape Concern Change from OL Baseline Endpoint | -0.44 [-0.57 to -0.31]
  Weight Concern Change from DB Baseline Endpoint | -1.47 [-1.63 to -1.31]
  Weight Concern Change from OL Baseline Endpoint | -0.53 [-0.66 to -0.39]

14. Secondary Outcome: Change in Eating Disorder Examination Questionnaire (EDE Q) Modified Global Score and Subscale Scores (Restraint, Shape, Concern, Weight Concern), and Items 4-6 Scores
Description: Eating Disorder Examination Questionnaire (EDE-Q) Modified global and subscale scores 4 subscale scores (Restraint, Eating Concern, Shape Concern, and Weight Concern) range from 0- 6, where 0 represents absence of the feature and 6 represents an extreme degree. An EDE-Q global score is calculated as average of 4 EDE-Q subscale scores.
  Item 4: Over the past 28 days, how many times have you eaten what other people would regard as an unusually large amount of food (given the circumstances)?
  Item 5: On how many of these times did you have a sense of having lost control over your eating (at the time that you were eating)?
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: events
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
events
  Item 4 Change from DB Baseline Endpoint | -17.4 [-18.2 to -16.6]
  Item 4 Change from OL Baseline Endpoint | -3.9 [-4.6 to -3.1]
  Item 5 Change from DB Baseline Endpoint | -16.6 [-17.4 to -15.8]
  Item 5 Change from OL Baseline Endpoint | -3.5 [-4.2 to -2.8]

15. Secondary Outcome: Change in Eating Disorder Examination Questionnaire (EDE Q) Modified Global Score and Subscale Scores (Restraint, Shape, Concern, Weight Concern), and Items 4-6 Scores
Description: Eating Disorder Examination Questionnaire (EDE-Q) Modified global and subscale scores 4 subscale scores (Restraint, Eating Concern, Shape Concern, and Weight Concern) range from 0- 6, where 0 represents absence of the feature and 6 represents an extreme degree. An EDE-Q global score is calculated as average of 4 EDE-Q subscale scores.
  Item 6: Over the past 28 days, on how many DAYS have such episodes of overeating occurred (i.e., you have eaten an unusually large amount of food and have had a sense of loss of control at the time)?
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: number of days
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
number of days
  Item 6 Change from DB Baseline Endpoint | -15.3 [-15.9 to -14.7]
  Item 6 Change from OL Baseline Endpoint | -3.3 [-3.8 to -2.7]

16. Secondary Outcome: Change in Binge Eating Clinical Global Impression-Severity (BE-CGI S) Score
Description: Binge-eating Clinical Global Impression-Severity (BE-CGI-S) The BE-CGI-S is a single value, clinician-rated assessment of illness severity, and 7-point scale with range from 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill subjects. A higher score is associated with greater illness severity.
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
units on a scale
  Change from DB Baseline Week 52 Endpoint | -2.7 [-2.8 to -2.6]
  Change from OL Baseline Week 52 Endpoint | -0.7 [-0.8 to -0.5]

17. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score and Subscale Scores (School/Work Disability, Social Life Disability, and Family Life Disability)
Description: The Sheehan Disability Scale (SDS) 3 subscales (work/school, social life, home life) are rated on the following scale: 0 = not at all; 1-3 = mildly; 4-6 = moderately; 7-9 =markedly; 10 = extremely. The 3 items can be combined into a single global measure of impairment (SDS total score) that ranges from 0 (unimpaired) to 30 (highly impaired). A higher subscale score and total score are associated with greater illness severity.
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
units on a scale
  Total Score Change from DB Baseline Endpoint | -8.2 [-9.0 to -7.4]
  Total Score Change from OL Baseline Endpoint | -1.5 [-2.1 to -0.9]
  Work/School Change from DB Baseline Endpoint | -2.0 [-2.3 to -1.8]
  Work/School Change from OL Baseline Endpoint | -0.4 [-0.6 to -0.2]
  Social Life Change from DB Baseline Endpoint | -3.2 [-3.5 to -2.9]
  Social Life Change from OL Baseline Endpoint | -0.5 [-0.7 to -0.3]
  Family Life Change from DB Baseline Endpoint | -2.9 [-3.2 to -2.6]
  Family Life Change from OL Baseline Endpoint | -0.4 [-0.6 to -0.2]

18. Secondary Outcome: Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score
Description: Hamilton Anxiety Rating Scale (HAM-A) total score HAM-A total score ranges from 0 to 56. A higher score is associated with a greater degree of anxiety.
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
units on a scale
  Change from DB Baseline Endpoint | 0.4 [0.0 to 0.9]
  Change from OL Baseline Endpoint | 0.6 [0.2 to 1.0]

19. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: Montgomery-Asberg Depression Rating Scale (MADRS) total score The MADRS total score ranges from 0 to 60, with higher scores indicating increased depressive symptoms
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dasotraline
Number analyzed (Participants) | 528
units on a scale
  Change from DB Baseline Endpoint | -0.6 [-1.1 to -0.1]
  Change from OL Baseline Endpoint | 0.4 [0.0 to 0.8]

20. Secondary Outcome: Change in SF-12 Two Component Scores (Physical, Mental Health)
Description: Change in SF-12 two component scores (physical, mental health) for Subjects Continued from Study SEP360-221 The SF-12 is a 12-item self-report questionnaire. Physical Component Summary (PCS) and Mental Component Summary (MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: Baseline, Week 52
Population: Safety
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Dasotraline
Number analyzed (Participants) | 204
units on a scale
  Mental Component Change from DB Baseline Endpoint | 1.25 [-0.44 to 2.95]
  Mental Component Change from OL Baseline Endpoint | -1.84 [-3.27 to -0.40]
  Physical Component Change from DB BL Endpoint | 2.56 [1.32 to 3.80]
  Physical Component Change from OL BL Endpoint | 0.87 [-0.16 to 1.90]

ADVERSE EVENTS:
Time Frame: An AE onset on or after the start of the open-label treatment period (treatment duration: 52 weeks) through 7 days after study drug discontinuation (14 days for serious adverse events and deaths)
Description: Treatment-emergent adverse events (TEAEs) are those reported adverse events with onset date on or after the first day of the open-label treatment period through 7 days after study drug discontinuation (14 days for serious adverse events and deaths).
Arm/Group | Dasotraline
All-Cause Mortality (participants affected / at risk) | 0/528
Serious Adverse Events (participants affected / at risk) | 21/528
Other Adverse Events (participants affected / at risk) | 295/528
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasotraline (N=528)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hemiplegic migraine (Nervous system disorders) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Substance-induced mood disorder (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasotraline (N=528)
Dry mouth (Gastrointestinal disorders) | 73 (81)
Nausea (Gastrointestinal disorders) | 27 (30)
Nasopharyngitis (Infections and infestations) | 30 (39)
Upper respiratory tract infection (Infections and infestations) | 51 (69)
Weight decreased (Investigations) | 77 (96)
Headache (Nervous system disorders) | 52 (60)
Anxiety (Psychiatric disorders) | 70 (77)
Insomnia (Psychiatric disorders) | 103 (114)
Irritability (Psychiatric disorders) | 27 (28)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT02684279/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT02684279/SAP_001.pdf